CLINICAL TRIAL: NCT01384812
Title: Headache Inducing Characteristics and Possible Changes in Cerebral Blood Flow After Administration of Prostaglandin E2 in Migraine Suffers Without Aura.
Brief Title: Prostaglandin E2 in Migraine Suffers Without Aura.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Troels Wienecke (Other)
Responsible Party: Sponsor-Investigator, Troels Wienecke, MD,PhD, Danish Headache Center
Organization: Danish Headache Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: DHC-PGE2-2011
Record Dates: First submitted 2011-06-20; First posted 2011-06-29 (Estimated); Last update posted 2011-11-09 (Estimated); Status verified 2011-11

CONDITIONS: "Migraine-like" Headache
MeSH Terms: interventions — Dinoprostone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Isoton sodium chloride (Placebo Comparator)
  Interventions: Drug: isoton sodium chloride
- Prostin E2 (dinoprostone) (Active Comparator)
  Interventions: Drug: dinoprostone

INTERVENTIONS:
Drug: dinoprostone — intravenous injection 0.4 μgr/kg/min for 25 min
  Other Names: Prostin E2
  Arms: Prostin E2 (dinoprostone)
Drug: isoton sodium chloride — intravenous injection for 25 min
  Other Names: placebo
  Arms: Isoton sodium chloride

SUMMARY:
The hypothesis of this study is that Prostaglandin E2 (PGE2) induces headache and dilatation of brain vessels in migraine patients without aura.

ELIGIBILITY:
Inclusion Criteria:

* Patients with migraine without aura

Exclusion Criteria:

* Tension type headache more than x 3 per month
* Other forms for primary headache
* Headache 24 h before the day of the investigation
* Migraine 48 h before the day of the investigation
* Hypertension
* Hypotension
* Pregnant/nursing
* Daily intake of medication (except oral contraceptives and migraine rescue medicine during migraine attack)
* Cardiovascular or central nervous system (CNS) disease
* Drug/alcohol abuse
* Psychiatric disease
* Asthma or any other lung diseases

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Headache score on a 10-point verbal rating scale (VRS). | 24 h
  Incidence of headache 0 indicated no headache; 1 indicated a different sensation, pounding or throbbing, but not necessarily painful; 5 indicated moderate headache and 10 indicated worst imaginable headache.

SECONDARY OUTCOMES:
Blood flow velocity in the middle cerebral artery (VMCA) measured by a Transcranial Doppler (TCD) ultrasonography (2MHz). | 90 min
  Changes from base line recorded every 10th min. until time 90 min on day 1 and day 2. The infusion takes 25 min from time 0.
Diameter of superficial temporal artery and radial artery measured by a high resolution ultrasound scanner, C-scan. | 90 min
  Changes from base line recorded every 10th min. until time 90 min on day 1 and day 2. The infusion takes 25 min from time 0.
Mean arterial blood pressure (MAP). | 90 min
  Changes from base line recorded every 10th min. until time 90 min on day 1 and day 2. The infusion takes 25 min from time 0.
Electrocardiography (ECG). | 90 min
  Changes from base line recorded every 10th min. until time 90 min on day 1 and day 2. The infusion takes 25 min from time 0.
Heart rate (HR). | 90 min
  Changes from base line recorded every 10th min. until time 90 min on day 1 and day 2. The infusion takes 25 min from time 0.
End-tidal partial pressure of pCO2 (PetCO2). | 90 min
  Changes from base line recorded every 10th min. until time 90 min on day 1 and day 2. The infusion takes 25 min from time 0.
Transcutaneous arterial oxygen saturation (SAT) | 90 min
  Changes from base line recorded every 10th min. until time 90 min on day 1 and day 2. The infusion takes 25 min from time 0.

CONTACTS AND LOCATIONS:
Overall Officials: Troels Wienecke, MD,PhD, Principal Investigator — Danish Headache Center
Locations (1):
- Danish Headache Center, Glostrup Municipality, Denmark